CLINICAL TRIAL: NCT01594788
Title: NGAL as a Marker of Acute Kidney Injury After Cardiac Surgery. Observational Study
Brief Title: Neutrophil Gelatinase-associated Lipocalin as a New Biomarker to Detect Acute Kidney Injury in Postoperative Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-NGL-2011-04
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-01

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Observational study aimed to test the ability of Neutrophil Gelatinase-associated Lipocalin (NGAL) concentration in blood and urine to predict and diagnose early acute renal failure (ARF) in patients after cardiac surgery with/without Cardiopulmonary bypass (CPB).

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18 years proposed for cardiac surgery with / without CPB.
* Accepting to participate in the study, with informed consent signed by the patient, guardian or family member.

Exclusion Criteria:

* Patients < 18 years.
* Patients do not agree to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalised patients
Sampling Method: Non-Probability Sample
Enrollment: 340
Dates: Start 2011-04; Study Completion 2012-12

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain